CLINICAL TRIAL: NCT04938791
Title: Relationship Between Perceive Effort, Physiological and Kinematic Changes During Upper Limbs Isometric Activity and Its Relationship With the Socio-demographic Characteristics
Brief Title: Fatigue and Kinematics During Isometric Activity of the Upper Limbs in Young and Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Escola Superior de Saude da Cruz Vermelha Portuguesa - Lisboa (Other)
Responsible Party: Principal Investigator, Helena Silva, Associate Senior Professor, Escola Superior de Saude da Cruz Vermelha Portuguesa - Lisboa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ESSCVP_FIS01/2021
Record Dates: First submitted 2021-06-04; First posted 2021-06-24 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Fatigue
Keywords: Respiration; Perceived; Kinematics; Performance
MeSH Terms: conditions — Fatigue; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Isometric activity (Experimental): All participants will be included in this arm
  Interventions: Other: Isometric activity

INTERVENTIONS:
Other: Isometric activity — Participants will do elevation of upper limbs and mantain a 90º degree flexion position in an unsupported way.
  Other Names: Isometric task

SUMMARY:
The aim of this study is to understand the relationship between perceived effort and physiological and kinematic variables caused by isometric activity of the upper limbs, as well as its relationship with socio-demographic characteristics, level of activity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Minimum age of 18 years;

Exclusion Criteria:

* Unable to provide written consent
* History of heart, cardiovascular and / or respiratory disease,
* Known untreated hypertension, cardiomyopathy, or exercise intolerance
* Presence of cognitive or neurological disorders
* Neuromuscular or orthopaedic disorder that limits the movement of the upper limb to 90° flexion or the maintenance of that position
* BMI ≥ 40

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in perceived effort on the Borg category-ratio 10-point scale (CR 10) | From baseline to end of activity, up to 15 minutes
  The perceived effort will be measured with Borg CR 10 scale. Possible scores range from 0 (no exertion at all) to 10 (extremely strong).
Change from Baseline in heart rate | From baseline to end of activity, up to 15 minutes
  Heart rate (heart beatings per minute) measured before and during activity to track cardiovascular changes during activity.
Change from Baseline in respiratory rate | From baseline to end of activity, up to 15 minutes
  Respiratory rate (respiratory cycles per minute) measured before and during activity to track changes in respiratory function during activity.
Change from Baseline in heart rate variability (HRV) | From baseline to end of activity, up to 15 minutes
  Interval (in milliseconds) between consecutive heartbeats measured before and during activity to track changes in autonomic function during activity.
Change from Baseline in electrodermal activity (EDA) | From baseline to end of activity, up to 15 minutes
  Electrical conductance (in microsiemens -µS) between two points of the hand over time measured before and during activity to track changes in autonomic function during activity.
Change from Baseline in muscle action potential amplitude through surface electromyography (sEMG) | From baseline to end of activity, up to 15 minutes
  Muscle action potential amplitude (in millivolts - ms) in surface electromyographic signal measured before and during activity to track muscular fatigue signs.
Change from Baseline in muscle action potential duration through surface electromyography (sEMG) | From baseline to end of activity, up to 15 minutes
  Muscle action potential duration (in milliseconds - ms) in surface electromyographic signal measured before and during activity to track muscular fatigue signs.
Change from Baseline in muscle action potential frequency through surface electromyography (sEMG) | From baseline to end of activity, up to 15 minutes
  Muscle action potential frequency (in hertz - Hz) of surface electromyographic signal measured before and during activity to track muscular fatigue signs.
Change from Baseline in respiratory pattern through inertial motion units (IMU) from baseline and during activity | From baseline to end of activity, up to 15 minutes
  Angular range of motion (in degrees) of rib cage and abdominal wall during upper limb activity measured before and during activity to track changes in respiratory pattern during activity
Change from Baseline in upper limb motion angular acceleration through inertial motion units (IMU) system | From baseline to end of activity, up to 15 minutes
  Angular acceleration (in m/s^2) of the arm measured before and during activity to track small movements of upper limb during isometric activity

SECONDARY OUTCOMES:
Health Status | Before isometric activity
  Health Status will be measured with Medical Outcomes Study (MOS) Short Form Health Survey 36 Item version 2 which measure health status of populations and individuals. Possible scores range from 0 0 (worst health status) to 100 (best health status).
Physical activity level | Before isometric activity
  Physical activity level will be measured using European Prospective Investigation into Cancer and Nutrition Physical Activity Questionnaire (EPIC-PAQ) that allows to estimate energy expenditure through self-report assessment of the intensity and average duration (per day, week and month) of physical activity performed by the participants in three distinct dimensions (professional, domestic and leisure).
  Participants are classified as ACTIVE if they perform: at least 150 minutes per week of moderate physical activity; OR at least 75 minutes per week of vigorous physical activity; OR at least 150 minutes per week of a combination of moderate-intensity activity. If they don't present any of the conditions described, they will be categorized as SEDENTARY.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel López López, PhD, Study Director — Universidade da Coruña
Locations (1):
- Escola Superior de Saúde da Cruz Vermelha Portuguesa - Lisboa, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Silva-Migueis H, Martinez-Jimenez EM, Casado-Hernandez I, Dias A, Monteiro AJ, Martins RB, Bernardes JM, Lopez-Lopez D, Gomez-Salgado J. Assessment and indicators of kinematic behavior and perceived fatigability. Rev Assoc Med Bras (1992). 2024 Feb 26;70(2):e20230924. doi: 10.1590/1806-9282.20230924. eCollection 2024. PMID 38422320